CLINICAL TRIAL: NCT03358953
Title: The Cardiovascular Impacts of Electronic Cigarettes to the Use of Nicotine Replacement Patches
Brief Title: The Cardiovascular Impacts of Electronic Cigarettes in Comparison to the Use of Nicotine Replacement Patches
Acronym: VAPOUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GN16CH051
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Smoking, Tobacco
Keywords: electronic cigarettes; cardiovascular; nicotine replacement patches
MeSH Terms: conditions — Tobacco Smoking; Vaping | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: E-cigarette versus nicotine replacement patches
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Cigarettes (Other): Participants wishing to quit tobacco smoking have an equal chance of being assigned to the electronic cigarette arm. They are supplied with a second generation e-cigarette to support their quit attempt with standard of care once weekly support sessions from NHS smoking cessation services.
  Interventions: Device: Electron Cigarette
- Nicotine replacement patches (Other): Participants wishing to quit tobacco smoking have an equal chance of being assigned to the nicotine replacement patch arm (standard care). They are supplied with a second generation e-cigarette to support their quit attempt with standard of care once weekly support sessions from NHS smoking cessation services.
  Interventions: Device: Nicotine Replacement Patch

INTERVENTIONS:
Device: Electron Cigarette — Blended Tobacco flavour, 18mg/ml
  Other Names: Smokemax Power e-cigarette
  Arms: Electronic Cigarettes
Device: Nicotine Replacement Patch — NiQuitin 21mg
  Other Names: NiQuitin
  Arms: Nicotine replacement patches

SUMMARY:
In Scotland tobacco-related illnesses account for in excess of 56,000 hospital admissions and a quarter of deaths each year. The resultant financial impact on NHS Scotland is over £300 million per annum. To minimise the clinical and financial burden of tobacco on national healthcare systems, Scotland's tobacco control strategy aims to create a "tobacco-free" generation by 2034, with the prevalence of smoking in the adult population reduced to ≤5 %. The multifaceted approach focuses upon tobacco prevention, protection and cessation.

In relation to smoking cessation, the use of EC has exponentially increased since 2011, and EC are presently the most popular nicotine replacement product used in England. The Public Health England (PHE) Report published in August 2015 advocates the use of EC when other smoking cessation aids have failed.

DETAILED DESCRIPTION:
Tobacco smoking (TS) remains a major health challenge for people in Scotland. EC are presently the most popular nicotine replacement product used in England. Recently NHS Greater Glasgow and Clyde (NHSGGC) have, like other Health Boards and Trusts in the UK, lifted the ban on ECs on hospital grounds. This decision has been based on recent evidence that ECs appear to be less harmful when compared to TS but it is acknowledged that the short- and long-term sequelae of ECs remain unknown. Systematic research focusing on the effectiveness of ECs on cardiovascular and pulmonary phenotypes is urgently needed.

The VAPOUR pilot study is a randomised control trial (RCT) investigating the short-term cardiorespiratory effects of EC in comparison to nicotine replacement patches (NRP) in smokers following 12 weeks of smoking cessation support with NHSGG&C Smokefree Community Services. We hypothesise that both EC and NRP users will experience improvements in cardiovascular and pulmonary function; but the effects may be less pronounced in EC users.

The data generated from the pilot study will be invaluable for sample size and power estimation towards the development of a larger scale study. If the data generated from such a trial demonstrate that EC have short-term cardiovascular and pulmonary health effects, this may reduce tobacco associated morbidity and mortality, improve patient care and minimise NHS healthcare costs, and lead to the development of long term studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years and wish to stop smoking. Smoker of at least 1-15 tobacco cigarette (TC) per day for ≥ six months Committed to attending weekly support sessions with NHSGGC Smokefree Services Must be willing to stop smoking tobacco cigarettes with the use of either nicotine replacement patches or an electronic cigarette with nicotine containing e-liquid.

Exclusion Criteria:

* Breastfeeding or pregnancy Use of EC or NRP within the past three months Uncontrolled hypertension - Blood pressure ≥165/95 mmHg

Established history of cardiovascular defined as:

Unstable angina, heart failure New York Heart Association (NYHA) Functional Classification classes III - IV Recent stroke, myocardial infarction, coronary artery bypass graft or percutaneous coronary angiogram within the last 3 months.

Established renal disease defined as eGFR <45 Established history of peripheral vascular disease Established history of Chronic Obstructive Pulmonary Disease. Illicit drug use Severe concurrent medical condition that would prevent participation in study procedures or malignant neoplasm or with life expectancy ≤ 3 months.

Major depressive illness or other psychiatric conditions. Participants who decline participation in the study or who are unable to provide informed consent

* History of allergies to active substances, excipients or delivery device (patch) in NRP or EC
* NRP: See current Summary of Product Characteristics
* EC: Nicotine, Propylene Glycol (PG), Glycerol and water.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-12-17 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function as assessed by flow mediated dilation | 12 weeks
  Change in endothelial function as assessed by flow mediated dilation

SECONDARY OUTCOMES:
Changes in respiratory function assessed through pulmonary function tests | 12 weeks
  Changes in respiratory function assessed through pulmonary function tests
Changes in endothelial function assessed by Endo-PAT2000, a non-invasive technique | 12 weeks
  Changes in endothelial function assessed by Endo-PAT2000, a non-invasive technique
• Changes in cardiovascular parameters through non-invasive haemodynamic measurements | 12 weeks
  • Changes in cardiovascular parameters through non-invasive haemodynamic measurements
• Changes in cardiovascular risk factor profile as assess through biomarkers markers of inflammation | 12 weeks
  • Changes in cardiovascular risk factor profile as assess through biomarkers markers of inflammation
• Changes in endothelial micoparticles | 12 weeks
  • Changes in endothelial micoparticles

CONTACTS AND LOCATIONS:
Overall Officials: Christian Delles, MBChB PhD, Study Chair — Glasgow University and NHS GGC
Locations (1):
- Glasgow Clinical Research Facility, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided